CLINICAL TRIAL: NCT01119781
Title: An Open-Label, Single-dose, Pharmacokinetic, Pharmacodynamic, and Safety Study of PEGylated Interferon Beta-1a (BIIB017) in Healthy Subjects and Subjects With Renal Impairment
Brief Title: A Single-Dose, Pharmacokinetic/Pharmacodynamic (PK/PD), & Safety Study of BIIB017 in Participants With Renal Impairment & Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 105RI101
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Healthy; Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- peginterferon beta-1a (Experimental): Single dose of peginterferon beta-1a at either 63 or 125 mcg in renal impaired Participants and healthy volunteers
  Interventions: Drug: BIIB017(peginterferon beta-1a)

INTERVENTIONS:
Drug: BIIB017(peginterferon beta-1a) — peginterferon beta-1a administered by a single subcutaneous (SC) injection using a pre-filled syringe on Day 1 at a dose of either 63 or 125 mcg depending on subpopulation assignment reflecting whether a healthy volunteer or level of renal impairment.

SUMMARY:
The primary objective of the study is to evaluate the pharmacokinetics (PK) of a single dose of PEGylated Interferon Beta-1a (BIIB017) administered subcutaneous in participants with renal impairment and in participants with normal renal function (healthy participants). A secondary objective of this study in this study population is to evaluate the safety and tolerability of a single dose of PEGylated Interferon Beta-1a administered subcutaneous.

DETAILED DESCRIPTION:
This study is an open-label, multicenter, non-randomized, serial-group study to estimate the effect of renal impairment on BIIB017 PK/PD. The study will be conducted at approximately 3 sites in the US and will enroll approximately 35 participants: 6 healthy volunteers (normal renal function), 9 with mild renal impairment, 6 with moderate renal impairment, 8 with severe renal impairment, and 6 participants with end stage renal disease who require hemodialysis 2 to 3 times a week.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects must have stable renal disease (i.e., no change in disease status within the last month) as determined by the Investigator with laboratory and clinical findings that support the diagnosis of renal impairment.
* Must have body mass index (BMI) between 18 and 35 kg/m2 inclusive.

Key Exclusion Criteria:

* History of any clinically unstable (in the past 6 months prior to screening) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, and psychiatric, or other major disease as determined by the Investigator.
* Any evidence of clinically significant findings on screening evaluations, which, in the opinion of the Investigator would pose a safety risk, or would interfere with appropriate interpretation of safety or PK data, or other unspecified reasons that, in the opinion of the Investigator or Biogen Idec, make the subject unsuitable for enrollment

NOTE: Other protocol defined Inclusion/Exclusion Criteria May Apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Area under the time-concentration curve (AUC) for serum concentrations of peginterferon beta-1a | Post-hemodialysis, pre-dose on Day 1, post dose at 6, 12, 24, 36, 48, 72, 96, 168, 240, 336, 408, 504, 576 and 672 hours

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Day 1 up to Week 5

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen

REFERENCES:
- [Derived] Hu X, Seddighzadeh A, Stecher S, Zhu Y, Goyal J, Matson M, Marbury T, Smith W, Nestorov I, Hung S. Pharmacokinetics, pharmacodynamics, and safety of peginterferon beta-1a in subjects with normal or impaired renal function. J Clin Pharmacol. 2015 Feb;55(2):179-88. doi: 10.1002/jcph.390. Epub 2014 Sep 23. PMID 25187030